CLINICAL TRIAL: NCT00160316
Title: Endometrial Safety of a Low Dose Continuous Combined 17 -Estradiol/Dydrogesterone Hormone Replacement Regimen (E2 0.5 mg/ D 2.5 mg) in Postmenopausal Women - A One-Year, Open Label, Multi-Center Study
Brief Title: Endometrial Safety Study of a 0.5 mg Estradiol and 2.5 mg Dydrogesterone Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Gregor Eibes, Solvay Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S102.3.117; 2004-000227-15
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Postmenopause
MeSH Terms: interventions — Estradiol; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 0.5 Mg Estradiol and 2.5 Mg Dydrogesterone

INTERVENTIONS:
Drug: 0.5 Mg Estradiol and 2.5 Mg Dydrogesterone — p.o. daily

SUMMARY:
The purpose of this study is to demonstrate endometrial safety of continuous combined 0.5 mg estradiol and 2.5 mg dydrogesterone.

ELIGIBILITY:
Inclusion Criteria:

* Amenorrhoea for >= 12 months.
* Serum estradiol and FSH level within the postmenopausal range
* Baseline endometrial biopsy assessed by light microscopic histological evaluation revealing: insufficient endometrial tissue for diagnosis because of insufficient available (atrophic) endometrial tissue (not because of an inaccessible cervix) and endometrial thickness < 5 mm (double layer) by transvaginal ultrasound, atrophic endometrium, secretory endometrium, menstrual type endometrium, proliferative endometrium

Exclusion Criteria:

* Previous systemic unopposed estrogen replacement therapy over 6 months or more.
* Any estrogen, progestogen, and/or androgen therapy in the last four weeks before Screening Visit (Visit 1). The baseline endometrial biopsy should in all cases be taken after cessation of the withdrawal bleeding due to previous hormone replacement therapy.
* History or presence of an estrogen dependent neoplasia (including breast- cancer).
* History or presence of malignant neoplasms other than basal or spinal cell carcinoma of the skin.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Presence of endometrial hyperplasia or a more serious endometrial outcome during the 52 week treatment period | 52 weeks

SECONDARY OUTCOMES:
Number of days with bleeding/spotting; Number of bleeding/spotting episodes; Number of days with a certain bleeding intensity (e.g. bleeding intensity =2); | 52 weeks
Length of bleeding free intervals; Amenorrhoea yes/no (absence of spotting and bleeding); Absence of bleeding yes/no; | 52 weeks
QualiPause Inventory (domains: psychological, vasomotor, somatic, sexual, menstrual, androgenic): average score of the single items within the domain; QualiPause Inventory 7D: weighted sum score of the symptoms | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (22):
- Croatia (4):
  - Site 10, Zagreb
  - Site 11, Zagreb
  - Site 12, Zagreb
  - Site 13, Zagreb
- Poland (7):
  - Site 32, Katowice
  - Site 30, Krakow
  - Site 35, Krakow
  - Site 36, Krakow
  - Site 34, Lublin
  - Site 31, Miechów
  - Site 33, Warsaw
- Romania (6):
  - Site 40, Bucharest
  - Site 41, Bucharest
  - Site 42, Bucharest
  - Site 43, Bucharest
  - Site 44, Bucharest
  - Site 45, Bucharest
- Ukraine (5):
  - Site 24, Donetsk
  - Site 20, Kiev
  - Site 21, Kiev
  - Site 22, Kiev
  - Site 23, Zaporizhzhya